CLINICAL TRIAL: NCT06091462
Title: The Effect of Virtual Reality Based Interactive Therapeutic Dementia Patient Education Program on the Knowledge, Attitude and Empathy Levels of Nursing Undergraduate Students
Brief Title: Virtual Reality and Nursing Students and Dementia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ayşe ARIKAN DÖNMEZ (Other)
Responsible Party: Sponsor-Investigator, Ayşe ARIKAN DÖNMEZ, associate professor, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-66777842-300-00003053868
Record Dates: First submitted 2023-09-18; First posted 2023-10-19 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Virtual Reality; Dementia; Education; Nursing Students
Keywords: Virtual Reality; Education; Nursing Students; dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality group (Experimental): Participants in the intervention group will log into the virtual reality-based interactive therapeutic patient education program with a username and password to be defined for them on the "hadi.hacettepe.edu.tr" website. After completing the dementia module in this program, the participants will complete the application by switching to the virtual reality-based interactive therapeutic patient education program.
  Interventions: Other: Virtual Reality Based Interactive Therapeutic Dementia Patient Education Program
- control group (No Intervention): Participants in the control group, on the other hand, will not receive any educational intervention other than standard education. In parallel with the completion of the application by the participants in the intervention group, the participants in the control group will complete the post-tests.

INTERVENTIONS:
Other: Virtual Reality Based Interactive Therapeutic Dementia Patient Education Program — Virtual reality is an interactive three-dimensional environment where computer simulation-based fictions and the real and virtual worlds are combined.
  Within the scope of this training, in the content of the module on the subject of Dementia; dementia definition, risk factors, signs and symptoms, complications, treatment and nursing care and patient and/or caregiver education. exists. After applying the dementia module, students complete the program by switching to a virtual reality-based simulation program for dementia.
  Arms: virtual reality group

SUMMARY:
SUBJECT: The Effect of Virtual Reality Based Interactive Therapeutic Dementia Patient Education Program on the Levels of Knowledge, Attitudes and Empathy towards Dementia OBJECTİVE: The research was planned to determine the effect of virtual reality-based interactive therapeutic dementia patient education program on the knowledge, attitude and empathy levels of nursing undergraduate students.

DESIGN: Pretest and posttest randomized controlled trial BACKGROUD:It is inevitable to strengthen and enrich nursing education with innovative teaching approaches in understanding the needs of individuals with dementia and informal caregivers and providing qualified nursing care for dementia, which is more difficult and intangible to understand compared to chronic diseases.From this point of view, it is expected that the virtual reality-based interactive therapeutic dementia patient education program to be implemented in this study will have positive ethics in the knowledge, attitude and empathy levels of nursing undergraduate students.

METHODS:

The research will be carried out between 16.10.2023 and 16.10.2024 with 50 second year nursing students from the faculty of nursing. Students will be divided into control and intervention groups of 25 people in the form of block randomization.Students in the intervention group will implement a virtual reality-based interactive therapeutic dementia patient education program.Students in the control group will not be given any program other than the routine education program.Both groups will be asked to fill simultaneously the dementia knowledge assessment scale, the dementia attitude scale, and the Jefferson empathy scale for nursing students before and after administration.Statistical analysis of the data will be made.

DETAILED DESCRIPTION:
PLACE OF RESEARCH The research was planned to be conducted at Hacettepe University Faculty of Nursing. As a result of the Research Infrastructure Project (No: TAY-2022-19754) supported by Hacettepe University Scientific Research Projects Coordination Unit, virtual reality simulation program is included in the infrastructure of the nursing faculty as of 2023. In this program, there are 3 different modular trainings on "Diabetes Mellitus", "Chemotherapy Treatment" and "Dementia" and simulation scenarios based on virtual reality for these subjects. The modular training and virtual reality-based simulation program is already active on the "hadi.hacettepe.edu.tr" website. Students who will benefit from this program can access the program after defining a user name and password. In the content of the module related to the subject of "Dementia" within the scope of this program; dementia definition, risk factors, signs and symptoms, complications, treatment and nursing care and patient and/or caregiver education. exists. After applying the dementia module, students complete the program by switching to a virtual reality-based simulation program for dementia.

THE UNIVERSE OF THE RESEARCH In the 2023-2024 academic year, Hacettepe University Faculty of Nursing will consist of 2nd year students. The main purpose of choosing this student group is that it is a group of students who have successfully completed the Basics of Nursing course in the 2nd year, have basic knowledge and skills in nursing care, but still do not have sufficient equipment in terms of intervening with the patient. While this student group was at the beginning of education and practices, it was thought that by determining the effect of the virtual reality-based interactive therapeutic dementia patient education program, it was thought that the use of this method in the further education processes would make significant contributions to the education of students.

SAMPLE OF THE RESEARCH G*Power- 3.1.9.4 software program was used to calculate the sample size and power of the research. The effect size was calculated as 0.85 based on the average score averages and standard deviations of the intervention and control groups towards dementia taken from a sample study. Accordingly, it was planned to complete the study with a total of 46 students, with 23 students in each group, at 80% power and 5% significance level, taking α=0.05 (Type I error). It is planned to complete the research with 50 students. Group intervention group (25 people) to be applied virtual reality; The group without any intervention (25 people) will be determined as the control group.

PREPARATİON OF DATA COLLECTİON FORM In the research, data will be collected with the following tools. PRE-TESTS include personal information form, Dementia Information Evaluation Scale, Dementia Attitude Scale and Jefferson Empathy Scale for Nursing Students; POST-TESTS include the Dementia Knowledge Assessment Scale, the Dementia Attitude Scale, and the Jefferson Empathy Scale for Nursing Students.

DATA COLLECTİON Students who meet the criteria for inclusion in the research and agree to participate in the research will be informed, and their questions regarding the operation of the research will be answered if they have any. It will be explained that the information collected in the interview will not be stated in the research and will not be published, and will be kept as a record. By explaining the Informed Voluntary Consent form, it will be ensured that they read the consent form and give their consent voluntarily, and it will be recorded. The data will be collected in forms and scales hand-delivered to the students by the researcher.

APPLİCATİON OF RESEARCH Students who meet the research criteria and agree to participate in the study will be given an acquaintance and information meeting before the research. Written informed consent will be obtained from students. After the participants to be included in the research are informed about the research face-to-face, they will be asked to fill out the Personal Information Form, Dementia Information Assessment Scale, Dementia Attitude Scale and Jefferson Empathy Scale for Nursing Students in order to complete the PRE-TESTS. After the completion of the Pre-Tests, the participants will be assigned to the intervention and control groups according to the block randomization method to be performed in a computerized environment.

INTERVENTION GROUP Participants in the intervention group will log into the virtual reality-based interactive therapeutic patient education program with a username and password to be defined for them on the "hadi.hacettepe.edu.tr" website. After completing the dementia module in this program, the participants will complete the application by switching to the virtual reality-based interactive therapeutic patient education program. After the participants complete the applications, it is planned to hold an analysis session for the training program. Immediately after the debriefing session is over, participants will be required to complete the POST-TESTS.

CONTROL GROUP Participants in the control group, on the other hand, will not receive any educational intervention other than standard education. In parallel with the completion of the application by the participants in the intervention group, the participants in the control group will complete the FINAL TESTS. Participants in the control group will be able to access the virtual reality-based interactive therapeutic dementia patient education program after the data and application of the study are completed.

EVALUATİON OF DATA The data to be obtained from the research will be evaluated by transferring them to the IBM SPSS (Statistical Packages for the Social Sciences) Statistics 23 program. While evaluating the data, descriptive statistics (mean, standard deviation, median, minimum, maximum) for continuous variables and frequency distribution for categorical variables will be used. Differences between categorical variables will be evaluated with Chi-square test and Fisher Exact test, and relations between numerical variables will be evaluated with Spearman Correlation Analysis. The conformity of the data to the normal distribution will be evaluated with the Shapiro Wilk test of normality and Q-Q graphs. Accordingly, if the parametric test assumptions are met, the Significance Test of the Difference Between Two Means in the comparison of independent group differences; If the parametric test assumptions cannot be met, the Mann-Whitney U test will be used. In dependent group comparisons, if parametric test assumptions are met, Analysis of Variance in Repeated Measurements and Significance Test of Difference Between Two Spouses; Friedman Test and Wilcoxon Paired Two Sample Test will be used when parametric test assumptions are not met. A p value of ≤0.05 will be considered statistically significant in all analyses.

ELIGIBILITY:
Inclusion Criteria:

* Being a second year student at Hacettepe Faculty of Nursing
* 18 years of age or older
* Voluntarily agree to participate in the study
* Have internet access
* Not having received a virtual reality-based training for dementia before

Exclusion Criteria:

* Not participating in any of the pretest-posttest tests
* Refusing to participate in the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-10-16 (Estimated); Primary Completion 2024-01-04 (Estimated); Study Completion 2024-10-16 (Estimated)

PRIMARY OUTCOMES:
Dementia Knowledge | Change from baseline scores at the end of 60 minutes.
  It assesses the level of dementia knowledge of health professionals, students and individuals.
  The scale consists of 17 items and is unidimensional. The lowest score is 0 and the highest score is 34. A higher score indicates that the participants have a higher level of knowledge about dementia. It will be applied to the students just before virtual reality simulation and after completing the training on the same day (each session is 60 minutes).
Dementia Attitude | Change from baseline scores at the end of 60 minutes.
  It measures attitudes towards dementia. The scale consists of 20 items in total and includes three dimensions: supportive, accepting and exclusionary attitudes. 6 items are reverse scored (2,6,8,9,9,16,17).
  Scores between 20-140 are obtained from the scale. The higher the score, the more supportive and accepting attitude increases, while exclusionary attitude decreases. It will be applied to the students just before virtual reality simulation and after completing the training on the same day (each session is 60 minutes). Change from baseline scores at the end of 60 minutes.
Jefferson Empathy Scale for Nursing Students | Change from baseline scores at the end of 60 minutes.
  The scale measuring empathy levels of nursing students consists of 20 items and 3 dimensions. Scores to be obtained from the scale 18-126 range. The higher the score, the higher the level of empathy. It will be applied to the students just before virtual reality simulation and after completing the training on the same day (each session is 60 minutes). Change from baseline scores at the end of 60 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)